CLINICAL TRIAL: NCT03059875
Title: Place of Comprehensive Geriatric Assessment (CGA) in Patients ≥ 75 Years Care, With Breast Cancer, After Screening With FOG (Oncology Geriatric Filter): Comparison Between CGA Before Surgery (Strategy A) vs. After Surgery (Strategy B)
Brief Title: Place of Comprehensive Geriatric Assessment in Patients ≥ 75 Years Care, With Breast Cancer, After Screening With FOG (Oncology Geriatric Filter)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GYNECO ONCOGER
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Surgery; 75 Years Old and More; Female Breast Cancer
Keywords: Breastcancer; Standardized Geriatric Evaluation; Onco-Geriatric Filter

ARMS (2):
- Strategy A (Other): Comprehensive Geriatric Assessment before the surgery of breast
  Interventions: Behavioral: Medical consultation for a Standardized Geriatric Evaluation
- Strategy B (Other): Comprehensive Geriatric Assessment after the surgery of breast
  Interventions: Behavioral: Medical consultation for a Standardized Geriatric Evaluation

INTERVENTIONS:
Behavioral: Medical consultation for a Standardized Geriatric Evaluation

SUMMARY:
The risk of diagnosis of cancer increases with age, especially breast cancer in elderly women. Elderly population is heterogeneous, regarding physiological reserves, comorbidities, disability and geriatric conditions. Comprehensive geriatric assessment (CGA) is a multidimensional approach to determine geriatric profile, in helping the therapeutic strategy. In-patients with diagnosis of cancer are screened with the FOG (oncology geriatric filter), to identify vulnerable subjects who may benefit from CGA. This scale of ten questions includes geriatric domains such as functional status, nutrition, mood, cognitive abilities and comorbidities. In elderly patients with breast cancer considered as fit (FOG=0), CGA is not necessary before adjuvant treatment. In vulnerable patients (FOG ≤ 1 and < 3), CGA is held in routine to discuss the adjuvant therapy feasibility. Patients with FOG ≥ 4 underwent CGA if palliative care is considered.

Patients in the intermediate group (FOG 1-3) are randomized to determine time of CGA, before or after surgery.

The aims of this study are to assess the outcomes regarding the time of CGA, in elderly female patients with breast cancer management, and to define the optimal place of CGA in care pathway.

ELIGIBILITY:
Inclusion Criteria:

* First breast cancer localized, indication of surgery
* Onco-geriatric filter (FOG) >= 1 ou < 4

Exclusion Criteria:

* Male, less of 75 years old
* Contraindication of surgery
* Breast cancer with metastasis
* Onco-geriatric filter (FOG) = 0 or 4

Min Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Compare Comprehensive Geriatric Assessment before the surgery and Comprehensive Geriatric Assessment after the surgery | 5 years

SECONDARY OUTCOMES:
Quality of life of patients | 5 years
  Questionnary EORTC QLQ - BR33
Patient satisfaction with their management | 5 years
  Questionnary REPERES 60 - Consumer Satisfaction Survey
Compare proportions of patients who received adjuvant chemotherapy and / or radiation standard | 5 years
Compare time to take care of Comprehensive Geriatric Assessment before the surgery and Comprehensive Geriatric Assessment after the surgery | 5 years
Compare the proportions of patients receiving adjuvant therapy, including complete hormone therapy | 5 years

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Hospital Center, Angoulême
  - Hospital center, Bressuire
  - Hospital Center, La Rochelle
  - Hospital center, Niort
  - University Hospital Center, Poitiers
  - Hospital center, Saintes